CLINICAL TRIAL: NCT02883114
Title: A Phase 1, Open-label, Two-period, Fixed-sequence Study To Estimate The Effects Of Multiple-dose Administration Of Itraconazole On The Single-dose Pharmacokinetics Of Pf-06648671 In Healthy Adults
Brief Title: An Open-Label, 2 Treatment Period,Study To Study The Drug Interaction Between Repeated Doses Of Itraconazole And Single Dose Pharmacokinetics (PK) Of PF-06648671 In Healthy Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Basic Science
Other Study IDs: B7991006
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
Keywords: PF-06648671; GSM; CYP3A; drug interaction
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single cohort (Experimental): single dose of PF-06648671 in period 1 and 14-day dose of itraconazole plus single dose of PF-06648671 in period 2
  Interventions: Drug: PF-06648671; Drug: Itraconazole

INTERVENTIONS:
Drug: PF-06648671 — Subjects will receive a single dose of PF-06648671 25 mg oral suspension on day 1 in period 1 and a single dose on Day 4 in period 2.
Drug: Itraconazole — Subjects will receive itraconazole 200 mg oral solution once a day for 14 days in period 2

SUMMARY:
This study is to evaluate the effect of multiple doses of itraconazole, the potent cytochrome P450 enzymes (CYP3A) inhibitor, on the pharmacokinetics of PF-06648671 following a single dose administration in healthy subject.

DETAILED DESCRIPTION:
Based on in vitro data, PF-06648671 was predominantly metabolized by CYP3A and therefore there is a potential risk that PF-06648671 PK will be affected by co-administered drugs that can inhibit CYP3A activity. This is a clinical drug interaction study to evaluate this potential drug interaction in human. In this study, healthy volunteers will take a single dose of 25 mg PF-06648671 in period 1 followed by at least 7 day washout. In period 2, same subjects will take 200 mg itraconazole oral solution once a day for 3 days, followed by co-administration of 200 mg oral solution and a single dose of 25 mg PF-06648671 on day 4 which are dosed approximately one hour apart with itraconazole is given first. The PF-06648671 PK will be collected 0-48 hours after dose in period 1 and 0-240 hrs in period 2. Safety will also be monitored throughout both periods.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and/or female subjects of non childbearing potential between the ages of 18 and 55 years at the time of screening, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG or clinical laboratory tests.
2. Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
4. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
2. Hypersensitivity or previous adverse events due to azole antifungals.
3. A positive urine drug testing.
4. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males within 6 months of Screening.
5. Use of tobacco or nicotine containing products in excess of the equivalent of 5 cigarettes per day.
6. Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study medication, whichever is longer.
7. Screening supine blood pressure >=140 mm Hg (systolic) or 90 mm Hg (diastolic), following at least 5 minutes of supine rest. If blood pressure (BP) is >=140 mm Hg (systolic) or 90 mm Hg (diastolic), the BP should be repeated two more times and the average of the three BP values should be used to determine the subject's eligibility.
8. Screening supine 12 lead ECG demonstrating corrected QT (QTc) >450 msec or a QRS interval >120 msec. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc or QRS values should be used to determine the subject's eligibility.
9. Subjects with ANY of the following abnormalities in clinical laboratory tests at Screening AND at Day 0, as assessed by the study specific laboratory and confirmed by a single repeat, if deemed necessary:

   * Aspartate aminotransferase (AST)/ serum glutamic oxaloacetic transaminase (SGOT) or alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) >1x upper limit of normal (ULN);
   * Total bilirubin>=1.5 x ULN; subjects with a history of Gilbert's syndrome may have a direct bilirubin measured and would be eligible for this study provided the direct bilirubin is ULN.
10. Fertile male subjects who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days, or longer based upon the compound's half life characteristics, after the last dose of investigational product.
11. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of investigational product. As an exception, acetaminophen/paracetamol may be used at doses of 1 g/day. Limited use of non prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case by case basis following approval by the sponsor.
12. History of hepatitis or positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (HBsAb), hepatitis B core antibody (HBcAb) or hepatitis C antibodies (HCV). As an exception, a positive HBsAb finding as a result of subject vaccination is permissible.
13. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
14. Unwilling or unable to comply with the Lifestyle Requirements described in this protocol.
15. Subjects who are investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
16. Any condition possibly affecting drug absorption.
17. Have any medical conditions, medical history, or are taking any medications that are contraindicated in the itraconazole prescribing information.
18. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Maximum Observed PF-06648671 Plasma Concentration (Cmax) | 0-48 hours in period 1 and 0-240 hours in period 2 following single dose PF-06648671
  Camx after single dose of 25 mg PF-06648671 in period 1 and period 2
Time to Reach Maximum Observed Plasma concentration (Tmax) | 0-48 hours in period 1 and 0-240 hours in period 2
  Tmax following single doses of PF-06648671 in period 1 and period 2
Area Under the Curve From Time Zero to Extrapolated Infinite Time in Plasma (AUCinf) | 0-48 hours in period 1 and 0-240 hours in period 2
  AUCinf following single doses of PF-06648671 in period 1 and period 2
Area Under the Curve from Time Zero to Last Quantifiable Plasma Concentration (AUClast) | 0-48 hours in period 1 and 0-240 hours in period 2
  AUClast following single doses of PF-06648671 in period 1 and period 2
Plasma Decay Half-life (t1/2) | 0-48 hours in period 1 and 0-240 hours in period 2
  t1/2 following single doses of PF-06648671 in period 1 and period 2
Apparent Oral Clearance (CL/F) | 0-48 hours in period 1 and 0-240 hours in period 2
  CL/F following single doses of PF-06648671 in period 1 and period 2
Apparent Volume of Distribution (Vz/F) | 0-48 hours in period 1 and 0-240 hours in period 2
  Vz/F following single doses of PF-06648671 in period 1 and period 2

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7991006&StudyName=A+Phase+1%2C+Open-label%2C+Two-period%2C+Fixed-sequence+Study+To+Estimate+The+Effects+Of+Multiple-dose+Administration+Of+Itraconazole+On+The+Single-dose+Pharmacokinetics+Of+Pf+06648671+In+Healthy+Adults
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7991006&StudyName=A+Phase+1%2C+Open-label%2C+Two-period%2C+Fixed-sequence+Study+To+Estimate+The+Effects+Of+Multiple-dose+Administration+Of+Itraconazole+On+The+Single-dose+Pharmacokinetics+Of+Pf-06648671+In+Healthy+Adults